CLINICAL TRIAL: NCT03831386
Title: The Impact of a Gravity Versus Vacuum Based Indwelling Tunneled Pleural Drainage System on Pain: A Multicenter, Randomized Trial
Brief Title: Gravity Versus Vacuum Based Indwelling Tunneled Pleural Drainage System
Acronym: NEWTON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Rocket Medical plc (Other); Swedish Medical Center (Other); Medical University of South Carolina (Other); University of Oxford (Other); Vanderbilt University Medical Center (Other); Northwest Community Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00158671
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vacuum (Active Comparator): The pleural fluid will be drained by the syringe system with a one-way valve tubing system provided in the kit. Selection of the vacuum pressure will be at the discretion of the proceduralist, as per standard of care. Participants in this arm will undergo Vacuum-Based IPC.
  Interventions: Procedure: Vacuum-Based IPC
- Gravity (Experimental): The pleural fluid will be drained using gravity drainage to a bag positioned at bedside. Participants in this arm will undergo Gravity-Based IPC.
  Interventions: Procedure: Gravity-Based IPC

INTERVENTIONS:
Procedure: Vacuum-Based IPC — An indwelling pleural catheter is placed inside the chest cavity to drain fluid from around the lungs. One end remains inside the body while the other drains via suction.
  Arms: Vacuum
Procedure: Gravity-Based IPC — An indwelling pleural catheter is placed inside the chest cavity to drain fluid from around the lungs. One end remains inside the body while the other drains via gravity.
  Arms: Gravity

SUMMARY:
Malignant pleural effusion remains a debilitating complication of end stage cancer, which can be greatly improved by the introduction of the indwelling tunneled pleural catheter (IPC). However, there is no standard of care regarding drainage and limited data on the utility of different drainage techniques. In addition, many patients develop discomfort and chest pain during drainage. The investigators propose to evaluate gravity drainage and suction drainage on quality of life measures and outcomes.

DETAILED DESCRIPTION:
Indwelling tunneled pleural catheters (IPCs) are used to alleviate pleural effusion as a first-line therapeutic (albeit palliative) intervention. Limited data currently exists on drainage techniques and the impact the techniques may have on quality of life. Current recommendations for IPC drainage range from daily drainage to once a week drainage, as well as only when needed for dyspnea. It has been theorized that active drainage of effusions may have an impact on the development of chest discomfort/pain, whereas passive regimens may allow for more gradual intrathoracic pleural changes and potentially offer a difference in drainage discomfort.

The objective of this investigation is to compare different drainage strategies of indwelling pleural catheters (IPCs) regarding patient quality of life and outcomes. Patients will undergo placement of a pleural catheter as per standard institutional protocol. Patients will be randomized on a 1:1 basis into the suction drainage (active) arm or the gravity drainage (passive) arm. Patients will receive follow-up at two weeks, four weeks, twelve weeks and then as needed post IPC placement per standard clinical protocol. All patients will be asked to fill out quality of life questionnaires and update drainage diary information with patient's providers.

Patients will undergo standard care treatment throughout the disease course and no different interventions regarding the pleural disease will be performed as a result of enrollment within this study. Study interventions/procedures will consist of questionnaires and patient self-reported documentation regarding patient's care and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indications for placement of IPC for malignant pleural effusion

  a. Pleural effusion with symptomatic improvement in dyspnea after drainage of ipsilateral effusion
* Clinically confident symptomatic malignant pleural effusion

  1. Histocytological proof of pleural malignancy
  2. Recurrent large pleural effusion in context of histologically proven cancer outside the pleural space
* Plans for placement of IPC within ten days of enrollment
* Age > 17 years
* Sufficient fluid on ultrasound to allow for safe insertion of IPC

Exclusion Criteria:

* Recent (less than 60 days) thoracic surgery or chest trauma causing chronic pain
* Pregnant or lactating mothers
* Previous ipsilateral chemical pleurodesis
* Current contralateral indwelling pleural catheter
* Known rib or thoracic skeletal metastasis causing pain
* Concern for active pleural infection
* Respiratory failure
* Irreversible bleeding diathesis
* Inability to provide care for indwelling tunneled pleural catheter
* Significantly loculated pleural space precluding drainage of pleural space, for which IPC alone will likely not offer symptomatic benefit
* Estimated life expectancy of < 30 days (however, active enrollment in hospice program is not an exclusion criteria)
* Inability to read/understand/write in the English language
* Inability to follow-up for appointments/protocol
* Subject has any clinical condition, diagnosis, or social circumstance that, in the opinion of the investigator would mean participation in the study would be contraindicated.
* Enrollment in alternative pleural catheter trial that would preclude enrollment within this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in chest pain as assessed by Visual Analog Scale (VAS) | Daily, up to 2 weeks
  The primary endpoint is the difference between the mean daily change in pain score during IPC drainage via the vacuum bottle technique and IPC drainage via the gravity bag technique over two weeks after IPC placement. Pre-drainage and post-drainage pain scores will be recorded each day of IPC placement. Measurements are in millimeters along a 10 cm VAS. VAS score is a range of 0 to 100. Lower limit is 0, meaning no pain; upper limit is 100, meaning extreme pain.

SECONDARY OUTCOMES:
Change in mean difference in chest pain as assessed by VAS | pre-IPC placement, 12 weeks post IPC placement or time of pleurodesis
  This secondary endpoint is the difference between the change in pain scores via vacuum bottle vs. gravity bag pre-IPC placement to the last available score after IPC placement. This last available score would be at 12 weeks or time of pleurodesis. Measurements are in millimeters along a 10 cm Visual Analog Scale (VAS). VAS score is a range of 0 to 100. Lower limit is 0, meaning no pain; upper limit is 100, meaning extreme pain.
Change in SF 36-Item Health Survey score | pre-IPC placement, 12 weeks post IPC placement or time of pleurodesis
  This secondary endpoint is the difference between SF 36-Item Health Survey 1.0 scores via vacuum bottle vs. gravity bag from pre-IPC drainage to last available score after IPC placement (at 12 weeks or time of pleurodesis). Scoring is a 2-step process in which the numerical response from the Survey is first converted into a 0-100 scale (0 as lowest and 100 as highest possible score) using a conversion table by SF developers. These new values would be averaged according to their group identified in a second conversion table.
Change in Functional Assessment of Chronic Illness Therapy (FACIT)-Dyspnea survey score | pre-IPC placement, 12 weeks post IPC placement or time of pleurodesis
  This secondary endpoint is the difference between FACIT-Dyspnea scores via vacuum bottle vs. gravity bag from pre-IPC drainage to the last available score after IPC placement (at 12 weeks or time of pleurodesis). Individual responses are converted into scores, then summed for an overall score. Scores range from 0 (lower limit) to 30 (high limit); the higher the score, the worse the dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, DO, Principal Investigator — Johns Hopkins University
Locations (6):
- United States (5):
  - Northwest Community Healthcare, Arlington Heights, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Swedish Medical Center, Seattle, Washington
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
De-identified individual study data will be used for analysis by lead PI and analyst. However, study is using REDCap database system with restrictions so that researchers only see individual data from their own site.